CLINICAL TRIAL: NCT05562245
Title: The Effect of Motivational Interviewing-Based Breastfeeding Education on Breastfeeding Motivation, Breastfeeding Success, and Breastfeeding Self-Efficacy Perceptions After Cesarean Section
Brief Title: Motivational Interviewing-Based Breastfeeding Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ebru Bekmezci, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/28
Record Dates: First submitted 2022-09-19; First posted 2022-09-30 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Breastfeeding; Motivation; Success; Self-Efficacy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The study was planned in a randomized controlled experimental design to evaluate the effect of motivational interviewing-based breastfeeding education on breastfeeding motivation, breastfeeding success and breastfeeding self-efficacy perception of primiparous mothers after cesarean section.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): 1. 1st hour after cesarean section Pre-tests and motivational interviewing-based breastfeeding education
  2. Postpartum 5-7th Day: When the mothers come to the hospital for control, a second motivational interviewing session will be held in the breastfeeding room and breastfeeding will be supported when necessary and a second measurement will be made.
  3. Postpartum 6th Week: The third motivational interviewing session will be held by going to the mothers' homes, breastfeeding will be supported when necessary and a third measurement will be made.
  4. Postpartum 3rd Month: In order to end the motivational interviewing, the fourth motivational interviewing session will be held by going to the mothers' homes and the fourth measurement will be made.
  Interventions: Other: Motivational Interviewing-Based Breastfeeding Education
- Control arm (No Intervention): 1st hour after cesarean section will be made pre-tests and routine breastfeeding training of the hospital will be given to mothers in the control group. Mothers will be followed up 5-7th days postpartum, postpartum 6th week, and postpartum 3rd month

INTERVENTIONS:
Other: Motivational Interviewing-Based Breastfeeding Education — Motivational interviewing is basically a directive and client-centered psychosocial intervention used to help individuals discover and analyze ambivalent emotions related to their health behaviors, to learn new skills and to improve their existing skills. One of the main guiding principles in motivational interviewing is self-support and empowerment. The interviews consist of one to four sessions lasting between 7.5-60 minutes.
  A total of four motivational interviews will be held with the mothers in the experimental group.
  Arms: Intervention arm

SUMMARY:
The general purpose of this project is; to evaluate effect of motivational interviewing-based breastfeeding education on breastfeeding motivation, breastfeeding success and breastfeeding self-efficacy perception of primiparous mothers after cesarean section.

The sub-aims of the study were to evaluate the effect of motivational interviewing-based breastfeeding education on breastfeeding outcomes of primiparous mothers who gave birth by cesarean section.

The study will be conducted between September 2022- March 2023 at Konya a private hospital.

DETAILED DESCRIPTION:
The research was planned as a randomized controlled experimental study. Block randomization method was used to determine the experimental and control groups. Randomization was done by a biostatistician outside the researcher. Mothers who meet the inclusion criteria and agree to participate in the study will be assigned to the experimental and control groups according to the randomization list.

A total of 80 primiparous mothers who gave birth by cesarean section, 40 in the experimental group and 40 in the control group, will be included in the study.

Pre-Test Information Collection Form at the 1st hour after Caesarean section, Postpartum 5-7. Day Follow-up Form, Postpartum 6th Week Follow-Up Form and Postpartum 3rd Month Follow-up Form, LATCH Breastfeeding Assessment Tool, Breastfeeding Self-Efficacy Short Form Scale, The Primipara Breastfeeding Motivation Scale, Confidence-sufficiency and importance a scale.

Breastfeeding education based on motivational interviewing will be held for mothers in the experimental group, 1st hour after cesarean section, 5-7th days postpartum, postpartum 6th week, and postpartum 3rd month. Routine breastfeeding training of the hospital will be given to mothers in the control group 1st hour after cesarean section and will be followed up 5-7th days postpartum, postpartum 6th week, and postpartum 3rd month. At the end of the study, the results of the mothers in the experimental and control groups will be evaluated.

The breastfeeding guide prepared by the researcher will be given to the mothers in the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study,
* Cesarean delivery,
* Does not have a condition that prevents breastfeeding,
* Married
* Primiparous,
* Not receiving general anesthesia,
* At least primary school graduate,
* 18 years and above,
* Do not have any chronic disease,
* The birth weight of the baby is 2500 g and above,
* Your baby's APGAR score is 7 and above in the 5th minute,
* Mothers whose babies do not have congenital and/or metabolic diseases will be included in the study.

Exclusion Criteria:

* Having multiple pregnancy and giving birth,
* Foreign nationals and do not speak Turkish,
* Having a history of preeclampsia, eclampsia and gestational diabetes,
* Mothers who develop complications during cesarean section and whose transfer to the service exceeds 1 hour (because breastfeeding will be delayed for the first hour),
* COVID-19 positive in the 1st hour after birth and having a condition that prevents breastfeeding,
* Those with a history of diagnosed mental or psychiatric illness will not be included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postpartum mothers
Enrollment: 76 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
LATCH Breastfeeding Assessment Tool | Change from LATCH Breastfeeding Assessment Tool at 3 months
  The scale consists of five evaluation criteria and each item is evaluated between 0-2 points. The score that can be obtained from the measurement tool can vary between 0-10.
Breastfeeding Self-Efficacy Short Form Scale | Change from Breastfeeding Self-Efficacy Short Form Scale at 3 months
  The scale consists of 33 items. It is scored between 1-5 and the lowest 14 and the highest 70 points can be obtained
The Primipara Breastfeeding Motivation Scale | Change from The Primipara Breastfeeding Motivation Scale at 3 months
  The Primipara Breastfeeding Motivation Scale: The scale consists of 29 items and is scored between 1-7. It has a total of four sub-dimensions. Evaluation is made by summing the scores obtained in each subgroup in the scale.
Confidence- sufficiency and importance a scale | Change from Confidence- sufficiency and importance a scale at 3 months
  It is a grading scale prepared in the form of a visual analog scale. The score that can be obtained from the scale varies in the range of 0-10 points.

SECONDARY OUTCOMES:
Rate of feeding the baby with only breast milk | 3 months
  1st hour after cesarean section, 5-7th days postpartum, postpartum 6th week, and postpartum 3rd month
Total breastfeeding time | 3 months
  1st hour after cesarean section, 5-7th days postpartum, postpartum 6th week, and postpartum 3rd month

CONTACTS AND LOCATIONS:
Overall Officials: Halime Esra Meram, PhD, Study Director — esrameran@selcuk.edu.tr
Locations (1):
- Medicana Konya Hospital, Konya, Turkey (Türkiye)